CLINICAL TRIAL: NCT05491954
Title: The Use of Continuous Glucose Monitors Among Women With Various Degrees of Glucose Intolerance: An Observational Cohort Study
Brief Title: Continuous Glucose Monitoring for Various Degrees of Glucose Intolerance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021H0009
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Diabetes, Gestational
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Glucose samples will be drawn
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (4):
- Euglycemic: Women who pass a 50g GCT with 1-hour glucose <135 mg/dL
  Interventions: Device: Dexcom G6
- Possible glucose intolerance: Women who fail a 50g GCT (1-hour glucose >135 mg/dL) and have 0/4 abnormal values on a 100g oral glucose tolerance test (OGTT) by Carpenter-Coustan values
  Interventions: Device: Dexcom G6
- Confirmed glucose intolerance: Women who fail a 50g GCT (1-hour glucose >135 mg/dL) and have 1/4 abnormal values on 100g GTT test by Carpenter-Coustan values
  Interventions: Device: Dexcom G6
- Gestational Diabetes Mellitus: Women who fail a 50g GCT (1-hour glucose >135 mg/dL) and have ≥2/4 abnormal values on 100g GTT test by Carpenter-Coustan values (Table 1), meeting criteria for GDM
  Interventions: Device: Dexcom G6

INTERVENTIONS:
Device: Dexcom G6 — Continuous glucose monitoring

SUMMARY:
Diabetes mellitus affects roughly 8% of pregnancies but is associated with significant perinatal and maternal morbidity, with 6% of pregnancies affected by gestational diabetes mellitus (GDM). Best practice guidelines recommend universal screening for gestational diabetes mellitus between 24-28 weeks of pregnancy in all women who do not have a diagnosis of pre-gestational diabetes mellitus. Among high-risk populations, performing an early diabetes screen is suggested at the initiation of prenatal care to evaluate for pre-gestational diabetes mellitus. Prior studies have demonstrated a difference in perinatal outcomes by comparing women with negative screening tests to those who fail a screen but pass a diagnostic test and those who are ultimately diagnosed with GDM. The investigators aim to use continuous glucose monitoring systems to study glycemic control in the early third trimester to further elucidate the differences between pregnant women with euglycemia, glucose intolerance, and GDM.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Women with a viable singleton or twin intrauterine pregnancy between 24 0/7 and 31 6/7 weeks gestation based on the best obstetric estimate by ACOG criteria
* Planning to deliver at OSU Wexner Medical Center
* Able to understand the study, and having understood, provide written informed consent in English

Exclusion Criteria:

* Abnormal early 50g GCT screen, thereby necessitating 100g OGTT at 24-28 weeks
* Known pregestational diabetes (type 1, type 2, MODY)
* 50g GCT >200 mg/dl leading to GDM diagnosis without the performance of 3hr 100g GTT
* Abnormal obstetrical ultrasound suspicious for major congenital abnormality
* Known or suspected fetal aneuploidy (by either CVS, amniocentesis, or cell-free DNA)
* Participation in another trial that may influence the primary outcome, without prior approval
* Participation in this trial in a prior pregnancy
* Higher order pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Women ages 18-45 living in central Ohio living with or without gestational diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Changes in glycemic control over late gestation as measured by A1c | 9 months
  Assessed by changes in glycemic control over late gestation as measured by HbA1c at the time of enrollment and delivery

SECONDARY OUTCOMES:
The number of neonatal hypoglycemic episodes | 1 week
  Assessed by requirement of neonatal antidiabetic care measured in the number of hypoglycemic episode requiring IV dextrose treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Buschur, MD, Principal Investigator — tOSU Medical Center
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be available to other researchers